CLINICAL TRIAL: NCT05905367
Title: Rapid IV Symptom-inhibited Fentanyl Induction (SIFI) to Facilitate Rotation Onto Oral Opioid Agonist Therapy (OAT)
Brief Title: Symptom-inhibited Fentanyl Induction
Acronym: SIFI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pouya Azar (Other)
Responsible Party: Sponsor-Investigator, Pouya Azar, Principal Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H23-00111
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use Disorder
Keywords: Fentanyl; Methadone; Morphine; Opioid agonist therapy
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Fentanyl; Methadone; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptom-inhibited IV fentanyl induction (Experimental): Symptom-inhibited IV fentanyl induction followed by opioid agonist therapy (OAT) with either oral methadone or slow-release oral morphine (SROM)
  Interventions: Drug: Fentanyl; Drug: Methadone; Drug: Slow-release oral morphine

INTERVENTIONS:
Drug: Fentanyl — Symptom-inhibited IV fentanyl induction
  Other Names: Fentanyl citrate; Fentanyl injection
Drug: Methadone — Opioid agonist therapy (OAT) with methadone at starting doses established by symptom-inhibited IV fentanyl induction
  Other Names: Methadone hydrochloride; Methadone oral product
Drug: Slow-release oral morphine — Opioid agonist therapy (OAT) with SROM at starting doses established by symptom-inhibited IV fentanyl induction
  Other Names: SROM; Kadian

SUMMARY:
The goal of this clinical trial is to test a treatment strategy for individuals with opioid use disorder (OUD) who use fentanyl. Participants will receive medically-administered doses of intravenous (IV) fentanyl at intervals until they are comfortable and do not have withdrawal symptoms. They then will be given opioid agonist therapy (OAT) once daily by mouth, which is the current standard treatment for OUD. In this trial, each participant's starting dose of OAT will be tailored to meet their opioid needs, based on the amount of IV fentanyl they received.

The main questions this trial aims to answer are:

* Is the IV fentanyl protocol feasible and safe for use in a community clinic setting?
* Will the protocol result in higher-than-standard starting doses of OAT? Are these doses safe, and will they enable participants to stay on OAT for a longer time?

DETAILED DESCRIPTION:
This is an open-label, single arm, prospective clinical trial involving 50 individuals with opioid use disorder (OUD) who use illicit fentanyl and for whom opioid agonist therapy (OAT) with either methadone or slow-release oral morphine (SROM) is clinically indicated. Participants who provide informed consent and are found to be eligible will undergo a "symptom-inhibited" fentanyl induction procedure under close medical supervision in a community clinic. A study doctor or nurse will administer intravenous (IV) fentanyl at 5-minute intervals until the participant indicates comfort and their opioid withdrawal symptoms are minimized, or until their sedation level is 2 on the Pasero Opioid-induced Sedation Scale (POSS). Immediately before the first dose of fentanyl, after each dose during the induction procedure, and every 5 minutes for 15 minutes (or until stable) after the final fentanyl dose, study staff will monitor the participants' level of sedation (POSS), withdrawal symptoms (Clinical Opiate Withdrawal Scale, COWS), and vital signs (heart rate, respiratory rate, blood pressure, oxygen saturation).

Selection of the appropriate OAT agent for each participant will be done in advance by the clinical addictions management team. Participants with a QTc interval >500 msec on screening ECG will not be eligible to receive methadone, and will be offered SROM if clinically appropriate. Participants with known chronic kidney disease will have serum creatinine tested for calculation of estimated glomerular filtration rate (eGFR) if they are to receive SROM; if eGFR is between 15 and 60 mL/min, SROM doses will be adjusted according to current recommendations [Lexicomp 2021]; if eGFR<15 mL/min, the participant will not be eligible to receive SROM.

The total cumulative dose of IV fentanyl administered during the induction phase (the loading dose) x 8 will be used as a proxy for the individual's 24-hour opioid tolerance, which in turn will be converted to oral morphine equivalents and used to calculate the appropriate starting dose of methadone or SROM, up to a maximum daily dose of 200 mg for methadone or 2000 mg for SROM. The first OAT dose will be administered under observation in the clinic, preferably on the same day and 15-30 minutes after the completion of the induction procedure. Participants will remain in the clinic under observation for 3 hours after the first dose of methadone or SROM. Vital signs, POSS, and COWS will be monitored before the first OAT dose, then hourly and prior to discharge. Study staff will assess the participants' satisfaction with the symptom-inhibited fentanyl induction process, using the single item Medication Satisfaction Questionnaire (MSQ) and 3-open ended questions. Participants will be discharged from the clinic when medically stable.

Participants will return to the study clinic once daily for 7 days for OAT dispensing and assessment of activity level in the previous 24 hours, vital signs, POSS, and COWS. An ECG will be performed on OAT Days 3 (+/- 2 days) and 7 (+/- 2 days) for participants receiving methadone. Methadone will be preferentially be maintained at the same dose for the first 7 days; however, methadone dose may be adjusted (up to a maximum daily dose of 200 mg) if felt to be safe and clinically indicated. SROM doses may be increased by 100 mg every 24-48 hours (consistent with current clinical guidelines from the British Columbia Centre on Substance Use) up to a maximum daily dose of 2000 mg if clinically indicated (presence of cravings or withdrawal symptoms, and absence of SROM-related adverse events and opioid toxicity).

After Day 7, OAT will be dispensed through a community pharmacy according to standard procedure. Participants will return to the study clinic for the following assessments at 7 days (up to +2 days) , 1 month (+/- 2 weeks), 3 months (+/- 1 month), 6 months (+/- 2 months), and 12 months (+/- 3 months) post-induction:

* Participant satisfaction with their current OUD treatment (single-item MSQ)
* Whether maintained on oral OAT and, if so, current dose
* Whether on prescribed opioids for risk mitigation, and if so, type and dose
* Self-reported illicit opioid use - type, route, amount, frequency
* Self-reported use of other substances - type, route, amount, frequency
* Withdrawal symptoms (COWS score)
* Urine drug test

At the same time points, additional information will be obtained from the clinic's electronic medical record (EMR) database:

* Overdose events requiring intervention (acute care or hospitalization)
* Hospitalizations, including diagnosis, route of admission, dates, duration
* Survival; if deceased, cause of death

ELIGIBILITY:
Inclusion Criteria:

1. Opioid use disorder (OUD) of any severity by DSM-5 Clinical Diagnostic criteria
2. Intentional use of unregulated fentanyl by any route (injection and/or inhalation) by participant self-report
3. Urine drug test (UDT) positive for fentanyl at screening or within 7 days prior to date of screening visit
4. Clinical indication to start OAT with methadone or SROM
5. Willing and able to provide written informed consent for study participation
6. If taking prescribed opioids for safer supply/risk mitigation, willing to discontinue them starting on study Day 1 and for the first 7 days of the study

Exclusion Criteria:

1. Individuals who are pregnant or breast-feeding
2. Currently receiving prescribed fentanyl in any form, e.g. fentanyl patch
3. Previous participation in this study
4. Current use of methadone >150mg/day or SROM >1300mg/day or buprenorphine extended-release in any dose
5. Use of buprenorphine-naloxone within the previous 3 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of clinically significant study drug-related adverse events requiring intervention | Count starting from the beginning of the IV fentanyl induction procedure up to the end of Day 7 on OAT
  Total number of clinically significant study drug-related adverse events (e.g. sedation, respiratory depression, hypoxia, QT prolongation) requiring intervention, occurring during the first week

SECONDARY OUTCOMES:
Starting doses of oral OAT | Immediately after IV fentanyl induction
  Starting doses of methadone or slow-release oral morphine (SROM)
OAT retention | Days 1-7 and 1, 3, 6, and 12 months after IV fentanyl induction
  Proportion of participants who are retained on OAT
Participant satisfaction with fentanyl induction | First 1 to 3 hours after IV fentanyl induction
  Qualitative interview and single-item Medication Satisfaction Questionnaire (MSQ)
Participant satisfaction with current OAT | Before IV fentanyl induction, and at Day 7 and 1, 3, 6, and 12 months after IV fentanyl induction
  Single-item MSQ
Withdrawal symptoms | Before, during, and during 1-3 hours after IV fentanyl induction; daily during first week on OAT; and at 1, 3, 6, and 12 months
  Clinical Opiate Withdrawal Scale (COWS) score
Overdose events | Day 7 and 1, 3, 6, and 12 months
  Opioid overdose events requiring Intervention (acute care or hospitalization)
Hospitalizations | Day 7 and 1, 3, 6, and 12 months
  Inpatient hospital admissions for any cause
Death | Day 7 and 1, 3, 6, and 12 months
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Azar, MD, Principal Investigator — University of British Columbia
Locations (1):
- Hope to Health Research & Innovation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Azar P, Ignaszewski MJ, Harris M, Barazanci Z, Davison R, Wong JSH, Maharaj A, Mathew N, Hall D, Guillemi SA, Foreman J, Barrios R, Montaner JSG. Rapid intravenous symptom-inhibiting fentanyl induction (SIFI) to optimize rotation onto oral opioid agonist therapy among individuals who use unregulated fentanyl: protocol for an open-label, single arm clinical trial. Addict Sci Clin Pract. 2025 Jul 29;20(1):58. doi: 10.1186/s13722-025-00586-7. PMID 40731024